CLINICAL TRIAL: NCT03043118
Title: A Pilot Study to Test the Influence of Vegetable Flavor Variety Using Herbs and Spices on Preschool Children's Vegetable Intake
Brief Title: Children's Taste Study to Increase Vegetable Intake in Preschoolers
Acronym: CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Assistant Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ChildrensTasteStudy
Record Dates: First submitted 2016-10-06; First posted 2017-02-03 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Obesity
Keywords: Eating Behaviors; Preschool; Vegetable Intake
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Variety (Experimental): Children receive three servings of vegetables each prepared with a different herb and spice blend.
  Interventions: Other: Variety Intervention
- No Variety - Control (No Intervention): Children receive three servings of vegetables each prepared with the same herb and spice blend.

INTERVENTIONS:
Other: Variety Intervention — Vegetable flavor variety created with multiple herb and spice blends
  Arms: Variety

SUMMARY:
Studies have shown that when exposed to a variety of food and flavor options people tend to consume more than when only one item is presented. This strategy has been used to increase vegetable intake in adults and during snacktime in children. Increasing vegetable consumption in children is important because higher vegetable intake has been associated with reduced risk of disease and because vegetables can help prevent weight gain by lowering the energy density of a meal. The purpose of this study was to investigate the effects of using herb and spice blends to create flavor variety in carrots as a model vegetable in a laboratory test meal. We predict that children will consume more vegetables and that the energy density of the meal will be lower when a variety of seasoned carrots are presented in comparison to a single flavor. A secondary goal of the study was to determine other influences that may predict children's liking and intake of seasoned vegetables, such as previous exposure, infant feeding practices, and genetic bitter sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of test meal foods
* Generally healthy

Exclusion Criteria:

* Food allergies
* Medications (prescription or OTC) that can affect taste, smell or appetite
* Medical conditions

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

PRIMARY OUTCOMES:
Chang in Vegetable Intake | Baseline and 1 week
  Consumption is measured by pre- and post- weights of carrot offered in both the variety and no variety conditions
Change in Total Food Intake | Baseline and 1 week
  Consumption is measured by pre- and post- weights of all meal items offered in both the variety and no variety conditions
Change in Meal Energy Density | Baseline and 1 week
  Calculated from the total calories consumed divided by the grams of food eaten

SECONDARY OUTCOMES:
Spice Intake Questionnaire | Baseline
  A survey of maternally reported herb and spice consumption during pregnancy and breastfeeding as well as current home use
Home Spice Checklist | Baseline
  A comprehensive checklist of 34 herbs and spices for parents to fill out at home to evaluate children's overall herb and spice exposure
Infant Feeding Practices | Baseline
  A survey of maternally reported feeding practices, include breastfeeding, formula feeding, and introduction to solid foods.
Liking of Broccoli with Herbs and Spices | Baseline
  Liking is measured using a child friendly 5-pt hedonic scale; pilot data for future studies looking to apply this technique to green vegetables
Liking of Carrots with Herb and Spice Blends | Baseline
  Liking is measured using a child friendly 5-pt hedonic scale

OTHER OUTCOMES:
Age | Baseline
  Age of the participant on visit 1
Height | Baseline
  Height measured in cm on a stadiometer
Weight | Baseline
  Weight measured to the 0.1 pounds using a digital scale
6-n-propylthiourcacil Sensitivity | Baseline
  Children switch and spit a 56 umol solution of 6-n-propylthiouracil and are classified as tasters if it described as "bitter" or "yucky" and non-tasters if it's described as "nothing" or "like water".
Body Mass Index | Baseline
  Calculated from height and weight (kg/m^2)
Children's Eating Behavior Questionnaire | Baseline
  A validated parent-reported questionnaire on children's typical eating behaviors and attitudes toward foods
Preschool Adjusted Liking Scale | Baseline
  A questionnaire to assess children's liking of various common foods and daily activities.
Family Demographics | Baseline
  A parent-reported questionnaire
Parental Feeding Practices | Baseline
  A parent-reported questionnaire on typical feeding practices

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Keller, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No